CLINICAL TRIAL: NCT03326492
Title: Evaluation of Anti-venoms Serum in Africa (ESAA). Data Collection in Real Life Conditions
Brief Title: Evaluation of Anti-venoms Serum in Africa
Acronym: ESAA
Status: Completed | Type: Observational
Sponsor: Institut Pasteur (Industry)
Collaborators: Cameroon Society of Epidemiology (CaSE) (Unknown); Centre International de Recherches d'Enseignements et de Soins (CIRES) (Unknown); Centre Pasteur du Cameroun (Other); Inosan Biopharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-092
Record Dates: First submitted 2017-08-29; First posted 2017-10-31 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2022-02

CONDITIONS: Snake Bites; Antivenins; Snake Venoms
Keywords: Snake bites; Antivenom serum; Snake venoms
MeSH Terms: conditions — Snake Bites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients bitten by a snake: Any patient over 5 years old going to a participating center for curative care following a snake bite.
  Participation to the study does not change usual follow-up of patients. Antivenom serum Inoserp Pan-Africa® injection will be decided according to the clinical evaluation of the patient.
  Interventions: Drug: Antivenom serum Inoserp Pan-Africa® injection

INTERVENTIONS:
Drug: Antivenom serum Inoserp Pan-Africa® injection — Participation to the study does not change usual follow-up of patients. All medical procedures will be performed and products will be used in a routine manner. Antivenom serum Inoserp Pan-Africa® injection will be decided according to the clinical evaluation of the patient.

SUMMARY:
There is little or no assessment under real-use conditions of the efficacy and the tolerance in the short, medium and long term of the antivenoms currently on the market and used in the treatment of snake bites.

The main objective is to assess the short term tolerance (< 2 hours post-injection) of the antivenom Inoserp Pan-Africa® (temporary market authorization) from Inosan laboratory currently available in Cameroon.

DETAILED DESCRIPTION:
Globally, the number of annual envenomings is estimated to be between 420,000 and 1,800,000. In sub-Saharan Africa, the annual number of envenomings is estimated at 315,000, leading to more than 9,000 amputations and about 7,000 deaths.

Snake bites are recognized by many authors as a neglected disease, whose incidence is underestimated or even unknown in several countries of sub-Saharan Africa. Few data are currently available on the morbidity, mortality and economic impact of snake bites.

In Cameroon and particularly in the northern part of the country, where the density of snakes is high, a few studies have been carried out. In 2002, the annual incidence of envenomings was estimated at 200/100 000 inhabitants, of which 85% was due to Echis ocellatus, and the lethality was 23.9% in some centers. The Ministry of Public Health introduced snake bites in 2015 as a priority health problem in the list of diseases being monitored. Thus, a national epidemiological surveillance system, with a weekly count of snake bites, has been implemented. In the first year, the incidence of annual snake bites was 11.4/100,000 inhabitants, representing more than 2,500 bites per year, including 43 deaths and a case fatality rate of up to 6% in some areas. The northern region (Adamaoua, North and Far North regions) (savanna and mixed zone) accounts for 40% of the country's burden and 77% of the deadly burden, while the forest zone accounts for 32% of the burden Morbid disease and 16% of the fatal burden (ministerial source). The monitoring is based on paper registers for bite reporting, supplemented by the sending of pharmacovigilance data by text messages, but this is very little used in current practice. The data collection system in Cameroon could therefore be improved in terms of both completeness and speed of centralizing data.

These estimates are likely to be well below the reality given the non-exhaustive nature of the data collection and the frequent use of traditional practitioners without referral in a hospital structure.

In recent years, FAV-Afrique® produced by Sanofi-Pasteur was the treatment of reference for venomous snake bites in West and Central Africa. It was the most evaluated and the most effective, reducing by a factor 5 to 10 the mortality. This anti-venom serum was polyspecific, containing an antivenom against ten species of snakes: Naja melanoleuca, nigricollis & haje; Dendroaspis polylepis, viridis & jamesoni, Bitis gabonica & arietans; Echis leucogaster & ocellatus.

However, Sanofi-Pasteur stopped production (last batch produced in January 2014 and expired in June 2016), making it necessary to use other snake antivenoms. Since the end of 2015, two new antivenoms are available in Cameroon where they are granted a provisional marketing authorization. Few clinical trials have evaluated the antivenoms currently available in Africa.

Some clinical efficacy and safety data have been published for Inoserp Pan-Africa®. However, the number of subjects was limited and assessment was limited to the period of hospitalization.

The lack of sufficient data on incidence and mortality associated with snake bites, the current weakness of the epidemiological data collection system and the presence on the market of antivenoms that are very little evaluated in terms of tolerance, effectiveness make action necessary.

The main objective of the study is therefore to assess the tolerance and the efficacy of the antivenom Inoserp Pan-Africa® from Inosan laboratory currently available in Cameroon.This study will be conducted under routine conditions in order to avoid bias in the results through the implementation of dedicated logistics which would not be representative of the usual conditions.

ELIGIBILITY:
Inclusion Criteria:

* Any patient over 5 years old (inclusive) visiting at a participating center for a snake bite with or without confirmed envenoming
* Informed consent to research

Exclusion Criteria:

* Patient refusal
* Under 5 year-old
* Antivenom serum administration before the arrival in the participating center
* History of severe allergic reactions to antivenom serum

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient over 5 years old (inclusive) visiting at a participating center for curative care following a snake bite, with or without confirmed envenoming, will be proposed to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 474 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Short term tolerance of the antivenom serum Inoserp Pan-Africa® | 30 months
  The short-term tolerance of the antivenom serum Inoserp Pan-Africa® will be assessed by the monitoring of the clinical signs occurence less than 2 hours post-injection

SECONDARY OUTCOMES:
Short term efficacy of the antivenom serum Inoserp Pan-Africa® | 30 months
  The short-term efficacy of the antivenom serum Inoserp Pan-Africa® will be assessed by the clinical evaluation when the patient arrives at the hospital and then regularly until 48 hours post-injection
Medium term tolerance of the antivenom serum Inoserp Pan-Africa® | 30 months
  The medium term tolerance of the antivenom serum Inoserp Pan-Africa® will be assessed by the monitoring of the clinical signs occurence more than 72 hours post-injection
Medium term efficacy of the antivenom serum Inoserp Pan-Africa® | 30 months
  The medium term efficacy of the antivenom serum Inoserp Pan-Africa® will be assessed by the vital status at 15 days of any patient who received at least one dose of the antivenom serum and by the reported consequences 15 days after the first dose administration of the antivenom serum

CONTACTS AND LOCATIONS:
Overall Officials: Armand Nkwescheu, MD, Principal Investigator — Cameroon Society of Epidemiology, Cameroon; Yap Boum, MD, Principal Investigator — Médecins Sans Frontière
Locations (13):
- Cameroon (13):
  - Hôpital de District d'Akonolinga, Akonolinga
  - Hôpital régional de Buea, Buea
  - Hôpital de District de Guider, Guider
  - Hôpital de District de Kolofata, Kolofata
  - Hôpital Régional de Limbe, Limbe
  - Hôpital de District de Mora, Mora
  - Hôpital Norvégien de N'Gaoundéré, N'Gaoundéré
  - Hôpital Régional de N'Gaoundéré, N'Gaoundéré
  - Hôpital Saint Malte de Njombe, Njombé
  - Hôpital de District de Poli, Poli
  - Hôpital de District de Sa'a, Sa'a
  - Hôpital de District de Tokombere, Tokonbéré
  - Centre des Urgences de Yaounde (CURY), Yaoundé

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chippaux JP, Amta P, Madec Y, Ntone R, Noel G, Clauteaux P, Boum Ii Y, Nkwescheu AS, Taieb F. Epidemiologic, clinical, and therapeutic aspects of formally identified Echis romani bites in northern Cameroon. PLoS Negl Trop Dis. 2025 Jul 28;19(7):e0013195. doi: 10.1371/journal.pntd.0013195. eCollection 2025 Jul. PMID 40720423
- [Result] Benhammou D, Chippaux JP, Ntone R, Madec Y, Amta P, Noel G, Karl FN, Perilhou A, Matchim L, Sanchez M, Ndifon M, Clauteaux P, Eteki L, Boum Y 2nd, Nkwescheu AS, Taieb F. Snakebites in Cameroon: Tolerance of a Snake Antivenom (Inoserp PAN-AFRICA) in Africa in Real-Life Conditions. Toxins (Basel). 2024 Mar 22;16(4):165. doi: 10.3390/toxins16040165. PMID 38668590
- [Result] Chippaux JP, Ntone R, Benhammou D, Madec Y, Noel G, Perilhou A, Karl F, Amta P, Sanchez M, Matchim L, Clauteaux P, Eteki L, Ndifon M, Boum Y, Nkwescheu AS, Taieb F. Real life condition evaluation of Inoserp PAN-AFRICA antivenom effectiveness in Cameroon. PLoS Negl Trop Dis. 2023 Nov 8;17(11):e0011707. doi: 10.1371/journal.pntd.0011707. eCollection 2023 Nov. PMID 37939111